CLINICAL TRIAL: NCT00061581
Title: Peripheral Blood Mobilized Hematopoietic Precursor Cell Transplantation Followed by T Cell Add-Back for Hematological Malignancies - Effect of Irradiated Donor Lymphocytes on Chimerism
Brief Title: Experimental Bone Marrow Transplant Protocol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030192; 03-H-0192; NCT00066300 (obsolete NCT alias)
Record Dates: First submitted 2003-05-29; First posted 2003-05-29 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2017-06-14

CONDITIONS: Acute Lymphocytic Leukemia; Chronic Myeloid Leukemia; Acute Myelocytic Leukemia; Myelodysplastic Syndromes; Myeloproliferative Disorders
Keywords: Chronic Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia (AML); Chronic Lymphocytic Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma; Graft-Versus Leukemia/Myeloma; Graft-Versus-Host Disease; Cyclosporine; Fludarabine; Myelodysplasia Syndrome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Neoplasms, Plasma Cell; Graft vs Host Disease

INTERVENTIONS:
Device: Isolex 300i Stem Cell Selection

SUMMARY:
Bone marrow transplantation (BMT) is a risky procedure. If doctors could reduce the complications, BMT would be safer to use for a wider range of conditions. The purposes of this study are

* to prevent graft rejection by increasing the amount of immunosuppression and by giving some lymphocytes from the donor before transplant;
* to prevent graft-versus-host disease (GVHD) by transplanting T-cell depleted stem cells;
* to improve the immune effect against residual leukemia by the add-back of donor lymphocytes before transplant and six or more weeks after transplant.

Beyond the standard transplant protocol, study participants will undergo additional procedures. First, along with total body irradiation, patients will receive two drugs (a high dose of cyclophosphamide and fludarabine) to suppress immunity and prevent rejection of the transplant. Second, four days before the transplant, patients will be given donor lymphocytes that have been irradiated to make them incapable of causing GVHD. On the day of the transplant, patients will receive an infusion of T-cell depleted bone marrow stem cells. Finally, patients will receive two doses of add-back donor T-cells (45 and 100 days post transplant) and the immunosuppressive drug cyclosporine starting on day 44 until about six months after transplant.

Study participants must be between the ages of 10 and 56 and have a family member who is a suitable stem cell donor match.

DETAILED DESCRIPTION:
Stem cell transplant studies carried out by the NHLBI BMT Unit have focused on approaches to optimize the stem cell and lymphocyte dose in order to improve transplant survival and increase the graft-vs.-leukemia effect. The aim is to create the transplant conditions that permit rapid donor immune recovery without causing graft-versus-host disease (GVHD) by using no post-transplant immunosuppression in conjunction with a transplant depleted of T cells to a fixed low dose, below the threshold known to be associated with GVHD.

We have found that the outcome from transplant is improved by controlling the stem cell (CD34+ cell) and T lymphocyte (CD3+ cell) dose. In the last study, in this series, we used the Nexell Isolex 300i system to obtain high CD34+ doses depleted of lymphocytes to a fixed CD3+ T cell dose of 2 x 10(4)/kg. The use of the cell separator and the monoclonal antibodies was covered by IDE 8139. The study measured the incidence of acute GVHD and used chimerism assays to determine the percentage of donor and recipient cells circulating at different time-points after transplant. We found that in the first six weeks donor T cell chimerism varied widely reaching 100% only in 10/22 patients. Thus the goal or rapid donor immune recovery was achievable only in about half the patients. Patients with mixed donor-recipient T cell populations are known to be at higher risk for late graft rejection and leukemic relapse after transplant. Therefore the achievement of full donor chimerism is an important therapeutic goal.

To improve donor T cell chimerism we will test whether the addition of irradiated donor lymphocytes during the preparative regimen of the transplant can increase the chance of achieving 100% donor T cell chimerism within six weeks of transplant. It is known that irradiated lymphocytes do not cause GVHD and that they can suppress residual host immunity, thus promoting donor lymphocyte engraftment. The end point of the study will be the proportion of patients achieving full donor chimerism six weeks after transplant. Apart from this addition of irradiated lymphocytes and some minor modifications, this protocol will be identical to the predecessor protocol 02-H-0111. This involves the continued use of the Isolex 300i cell separator and the monoclonal antibodies provided by CTEP (anti CD 6, anti CD2, anti CD7). This is covered by a continuing IND for the selection of CD34+ and CD3+ cells for T cell depleted peripheral blood stem cell transplantation.

ELIGIBILITY:
* INCLUSION CRITERIA FOR RECIPIENTS:

Recipient

Ages 10-55 years inclusive (but less than 56)

Chronic myelogenous leukemia in chronic phase

A) Patients not treated with STI 571 under the age of 41 (subject to regular DSMB review).

B) 10-55 age limits patients in chronic phase who have failed treatment with STI-571.

C) 10-55 age limits patients in accelerated phase or blast transformation.

Acute lymphoblastic leukemia, any of these categories: Adults (greater than 18 years) in first remission with high-risk features (presenting leukocyte count greater than 100,000/cu mm, Karyotypes t9; 22, t4, t19, t11, biphenotypic leukemia) All second or subsequent remissions, primary induction failure, partially responding or untreated relapse.

Acute myelogenous leukemia (AML): AML in first remission Except AML with good risk karyotypes: AML M3 (t15; 17), AML M4Eo (inv 16), AML t (8; 21). All AML in second or subsequent remission, primary induction failure and resistant relapse.

Myelodysplastic syndromes, any of these categories: refractory anemia with transfusion dependence, refractory anemia with excess of blasts, transformation to acute leukemia, chronic myelomonocytic leukemia.

Myeloproliferative disorders (myelofibrosis, polycythemia vera, essential thrombocythemia) in transformation to acute leukemia

Chronic lymphocytic leukemia refractory to fludarabine treatment and with bulky progressive disease or with thrombocytopenia (less than or equal to 100,000/ml) or anemia (less than or equal to 10g/dl) not due to recent chemotherapy.

Non-Hodgkin s lymphoma including Mantle cell lymphoma relapsing or refractory to current chemotherapy and monoclonal antibody treatment and unsuitable for autologous stem cell transplantation.

No major organ dysfunction precluding transplantation.

DLCO greater than or equal to 60% predicted.

Left ventricular ejection fraction: greater than or equal to 40% predicted.

ECOG performance status of 0 or 1.

For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: Written informed consent from one parent or guardian. Informed oral consent from minors: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

Negative pregnancy test for women of childbearing age.

INCLUSION CRITERIA FOR DONORS:

HLA 6/6 identical family donor

Weight greater than or equal to 18 kg

Age greater than or equal to 2 or less than or equal to 80 years old

Fit to receive G-CSF and give peripheral blood stem cells (normal blood count, normotensive, no history of stroke)

For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: Written informed consent from one parent or guardian and informed assent: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

EXCLUSION CRITERIA FOR RECIPIENTS (any of the following):

Patient pregnant

Age less than 10 years and 56 years or more

Patients with CML in chronic phase who are 41 years or over in whom STI 571 is the treatment of choice

ECOG performance status of 2 or more

Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the BMT treatment unlikely, and making informed consent impossible.

Major anticipated illness or organ failure incompatible with survival from BMT

DLCO less than 60% predicted.

Left ventricular ejection fraction: less than 40% predicted

Serum creatinine greater than 3mg/dl

Serum bilirubin greater than 4 mg/dl

Transaminases greater than 3 times the upper limit of normal

HIV positive

History of other malignancies except basal cell or squamous carcinoma of the skin, positive PAP smear and subsequent negative follow up, individuals with diseases listed in eligibility criteria for this protocol, but where debility or age makes the risk of intensive myeloablative therapy unacceptable. This includes patients who have received busulfan treatment for more than 6 months continuously. These patients will be considered for a non-myeloablative allogeneic transplantation protocols.

EXCLUSION CRITERIA:

Donor (any of the following)

Pregnant or lactating

Donor unfit to receive G-CSF and undergo apheresis. (Uncontrolled hypertension, history of congestive heart failure or unstable angina, thrombocytopenia)

HIV positive. Donors who are positive for HBV, HCV or HTLV-1 may be used if the risk-benefit ratio is considered acceptable by the patient and investigator.

Weight less than 18 kg

Age less than 2 or greater than 80 years

Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the BMT treatment unlikely, and making informed consent impossible

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2003-05-19; Primary Completion 2007-12-28 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Acute and chronic graft-versus-host disease, transplant-related mortality (TRM), overall mortality, leukemic relapse, CMV reactivation and disease, and graft failure.

CONTACTS AND LOCATIONS:
Overall Officials: A. John Barrett, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Couriel D, Canosa J, Engler H, Collins A, Dunbar C, Barrett AJ. Early reactivation of cytomegalovirus and high risk of interstitial pneumonitis following T-depleted BMT for adults with hematological malignancies. Bone Marrow Transplant. 1996 Aug;18(2):347-53. PMID 8864445
- [Background] Mavroudis D, Read E, Cottler-Fox M, Couriel D, Molldrem J, Carter C, Yu M, Dunbar C, Barrett J. CD34+ cell dose predicts survival, posttransplant morbidity, and rate of hematologic recovery after allogeneic marrow transplants for hematologic malignancies. Blood. 1996 Oct 15;88(8):3223-9. PMID 8874224
- [Background] Mavroudis DA, Read EJ, Molldrem J, Raptis A, Plante M, Carter CS, Phang S, Dunbar CE, Barrett AJ. T cell-depleted granulocyte colony-stimulating factor (G-CSF) modified allogenic bone marrow transplantation for hematological malignancy improves graft CD34+ cell content but is associated with delayed pancytopenia. Bone Marrow Transplant. 1998 Mar;21(5):431-40. doi: 10.1038/sj.bmt.1701120. PMID 9535034
- [Derived] McIver ZA, Yin F, Hughes T, Battiwalla M, Ito S, Koklanaris E, Haggerty J, Hensel NF, Barrett AJ. Second hematopoietic SCT for leukemia relapsing after myeloablative T cell-depleted transplants does not prolong survival. Bone Marrow Transplant. 2013 Sep;48(9):1192-7. doi: 10.1038/bmt.2013.39. Epub 2013 Mar 25. PMID 23524640
- [Derived] McIver Z, Melenhorst JJ, Wu C, Grim A, Ito S, Cho I, Hensel N, Battiwalla M, Barrett AJ. Donor lymphocyte count and thymic activity predict lymphocyte recovery and outcomes after matched-sibling hematopoietic stem cell transplant. Haematologica. 2013 Mar;98(3):346-52. doi: 10.3324/haematol.2012.072991. Epub 2012 Oct 12. PMID 23065508